CLINICAL TRIAL: NCT06097741
Title: Pulmonary MRI Using Ultra Short /Zero TE Sequences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Mareen Kraus, Principal Investigator, IWK Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1029785
Record Dates: First submitted 2023-10-13; First posted 2023-10-24 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2024-10

CONDITIONS: Image
Keywords: Magnetic Resonance Imaging; Sequences

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MRI sequence (Other): patients receive an MRI
  Interventions: Device: MRI sequences

INTERVENTIONS:
Device: MRI sequences — Ultra short / zero TE sequence on MRI being tested on healthy patients and improved by manually fine tuning the sequence

SUMMARY:
Modern imaging modalities, especially magnetic resonance imaging (MRI) have greatly advanced in recent years. Through technical advances, proton-based magnetic resonance imaging (MRI) has steadily increased in use to assess pulmonary structures in the pediatric population especially in Europe. Such technical developments have advanced by overcoming rapid decaying of transverse relaxation time and cardiac/chest movement synchronization, showing MRI to be feasible with respect to morphological and functional assessment of pulmonary impairment, in chronic lung disease such as cystic fibrosis for disease progression and prediction of exacerbation. However pulmonary imaging with MRI has also been feasible to detect pulmonary nodules in malignancies (allowing for spatial resolution).

DETAILED DESCRIPTION:
This prospective study will enable developing/ fine tuning for an optimized ultra-short echo/zero echo MRI sequence to enable pulmonary imaging with assessment of detailed lung structures which is important in patient with chronic lung disease. This will enable radiation sparing through x-ray and computed tomography, especially reduce the accumulation dose in long term follow up imaging of patients with chronic lung disease. Also, detailed pulmonary imaging enables more detailed imaging in comparison to the standard reference of care often using radiographs, can pick up disease prior to clinical symptoms, is a useful tool to assess treatment outcome and can sometimes even prevent chronic changes by early disease diagnosis and rapid treatment. This is of particular interest in patients with chronic lung disease, such as cystic fibrosis, but also other congenital lung diseases such as congenital pulmonary airway malformation (CPAM) or malignant diseases which will otherwise have a second CT imaging to assess the lung.

The investigators will recruit healthy volunteers to assess the available MR sequences on the 1.5 T MRI scanner at the IWK health Centre in the Department of Diagnostic Imaging and either fine tune/modify the existing protocol with the help of the MRI technologist and application specialists or build a new sequence according to the most recent literature. The aim is to recruit 15 patients of different age group (aged 3- 18 years old) to assure a robust imaging protocol for all age groups. Especially, the preschool age group can be more challenging due to increased cardiac and respiratory motion, but also the understanding of the diagnostic imaging with guidance of the in house child life support as well as parental guidance and support, the possibility to watch a video on the MRI scanner to distract the patient as best as possible since the aim is to conduct the short pulmonary MRI protocol without the need for sedation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants (without prior history of pulmonary disease)
* Ages 3 - 18 years old

Exclusion Criteria:

* prior history of pulmonary disease
* implants
* surgeries
* pregnancy
* metal devices
* braces
* anything that would exclude them from taking an MRI

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Image Quality | Image acquisition in November will undergo immediate assessment to potentially enhance imaging quality. Images will then be promptly reviewed on PACS after acquisition and post-trial termination, with parameters compared for an optimal sequence protocol.
  Imaging acquisition with and without breath hold is being tested and ultimately reconstruction of the acquired imaging. It will be assessed if the imaging is going to be of clinical and diagnostic standard by an experienced pediatric and pulmonary radiologist who has worked with ultra-short/zero TE sequences in clinical routine before. Here by imaging will be assessed looking at overall quality, signal, movement artifact of heart and breathing. Feasibility of preschool children to undergo imaging protocol in terms of protocol length, breathing maneuvers, general tolerability.
Acquisition Time | Volunteers get a call for MRI details. After 3 days, if they agree, we set imaging appointments. The PI and tech clarify, perform imaging, confirm post-exam well-being, and have a brief follow-up chat.
  The image acquisition is meant to take place in November and imaging will be assessed at the time of acquisition so that alteration of imaging parameters might improve imaging overall. The images itself will again be viewed on PACS shortly after acquisition and after termination of the trial imaging acquisition. Parameters will be compared to elaborate the best possible sequence protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Mareen Kraus, MD, Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No